CLINICAL TRIAL: NCT02040467
Title: Registry for Proton Beam Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201209025
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal is to collect information on each patient treated with proton beam radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

-Any patient receiving proton beam therapy is eligible for enrollment to this registry (regardless of diagnosis, age, other concurrent therapies, etc.) provided s/he consents to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient receiving proton beam therapy
Sampling Method: Non-Probability Sample
Enrollment: 1243 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Treatment-specific data for all patients receiving proton beam radiation therapy | 10 years
  Treatment-specific data collection record for all patients receiving proton beam radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Michalski, M.D., Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers University, New Brunswick, New Jersey
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu